CLINICAL TRIAL: NCT03654131
Title: Stereotactic Body Radiation Therapy vs. Microwave Ablation for Colorectal Cancer Patients With Metastatic Disease in the Liver - a Randomized Phase II Trail
Brief Title: Microwave Ablation Versus Stereotactic Body Radiotherapy for Colorectal Liver Metastases in Oligometastatic Disease: a Prospective, Randomised, Phase 2 Trial
Acronym: LAVA-CRLM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Signe Lenora Risumlund, Senior consultant, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-18000085
Record Dates: First submitted 2018-08-27; First posted 2018-08-31 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Carcinoma; Liver Metastases
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: SBRT for oligometastases in the liver from colorectal cancer patients. Standard considered MWA.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MWA (Active Comparator): Percutaneous ultrasound-guided MWA or open surgery MWA. The patient is fully anesthetized during the treatment.
  Interventions: Device: MWA
- SBRT (Active Comparator): 3 fractions of 15 Gy (in total 45 Gy), 3 fractions per week. The dose is prescribed to the PTV encompassing 67% isodose. The SBRT plan is normalized such that the mean dose to the GTV is 100% = 67.5 Gy.
  Interventions: Radiation: SBRT

INTERVENTIONS:
Device: MWA — Patients are allocated to one of the two arms in a 1:1 randomization
  Arms: MWA
Radiation: SBRT — Patients are allocated to one of the two arms in a 1:1 randomization
  Arms: SBRT

SUMMARY:
The LAVA-CRLM trial (Local Ablation Versus Ablative radiotherapy in ColoRectal Liver Metastases) is a prospective, randomised, phase 2 study designed to compare local control and safety of microwave ablation (MWA) versus stereotactic body radiotherapy (SBRT)in patients with colorectal liver metastases and oligometastatic disease. Primary endpoint is freedom form local lesion progression.

DETAILED DESCRIPTION:
Colorectal cancer patients with 1-3 liver metastases (diameter ≤4.0 cm) found unsuitable for resection are randomized 1:1 to either MWA or SBRT. Chemotherapy is allowed. Curative treatment of extrahepatic disease must be initiated in patients with lung metastases and/or primary tumors. Patients will be analyzed according to the intention-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

1. Colorectal cancer patients with oligo metastatic disease in the liver (1 to 3 tumors), and where metastases are found unsuitable for resection because of

   1. non-resectability
   2. small metastasis localized deep in the liver, where a parenchyma sparing intervention is preferred over an extensive resection
   3. previous extensive liver surgery
   4. comorbidity
2. The multidisciplinary team should all agree that both percutaneous or open surgical MW-ablation and SBRT are safe as first treatment choice for the individual patient.
3. Tumor sizes ≤4.0 cm
4. Age > 18 years
5. Signed informed consent

Exclusion Criteria:

1. Previous radiotherapy to the liver
2. Liver volume < 700 ml
3. Another active cancer disease within the past 36 months
4. Not able to understand written or oral protocol information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2027-12-03 (Estimated); Study Completion 2029-12-03 (Estimated)

PRIMARY OUTCOMES:
Freedom from local lesion progression (analyzed on patient-level) | 1 year
  * Defined as the time from randomization to local progression
  * Censoring: death from any cause, last follow-up
  * No censoring on disease progression outside of the treated lesions
  * Local lesion progression is defined as >20% increase in the longest diameter and minimum 5 mm increase talking as reference the smallest longest diameter recorded since the treatment started in any of the treated lesions

SECONDARY OUTCOMES:
Overall survival | From enrollment to 01/01/2026 - minimum follow-up 1 year after treatment for all randomised patients.
  * Defined as the time from randomization to death from any cause
  * Censoring: last follow-up
≥ grade 3 toxicity potentially associated with the treatment | 1 month after treatment
  - Using the Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Toxicity profile as descriptive statistics | From enrollment to last follow-up 5 years after treatment
  Using the Common Terminology Criteria for Adverse Events (CTCAE) v 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Righospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available upon reasonable request to the corresponding author after publication of all analyses of the primary and secondary trial endpoints
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication of all analyses of the primary and secondary trial endpoints and until 5 years after.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose for individual participant data meta-analysis. For this please contact the principal investigator of the trial. Data sharing will be conducted in accordance with Danish law on the processing of personal data, regulations of the Danish Data Protection Authority, and applicable health legislation.
  Contact Principal investigator Signe Lenora Risumlund Senior Oncologist Department of Oncology, Blegdamsvej 9, 2100 Copenhagen, Capital Region of Denmark, Denmark Signe.lenora.risumlund@regionh.dk
URL: https://clinicaltrials.gov/study/NCT03654131

DOCUMENTS (2):
  • Study Protocol (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/31/NCT03654131/Prot_002.pdf
  • Statistical Analysis Plan (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/31/NCT03654131/SAP_003.pdf